CLINICAL TRIAL: NCT03854136
Title: Treatment and Complications of Musculoskeletal Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Moiz Ali, Research Volunteer, Aga Khan University
Other Study IDs: AKU
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Musculoskeletal Diseases or Conditions
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Excision of tumor — Wide margin excision of tumors +/- limb preservation

SUMMARY:
Patients being treated for musculoskeletal tumors were included in the study. Their records were reviewed retrospectively and data was gathered regarding types of surgeries and post-operative complications including recurrence or development of secondary tumors if any.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing treatment for musculoskeletal tumors

Exclusion Criteria:

* Patients who did not undergo any surgical intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages and gender who underwent surgical intervention for musculoskeletal tumors at our institution were included
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 1995-07 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 5 years
  Recurrence of tumor at primary site

CONTACTS AND LOCATIONS:
Overall Officials: Obada Hassan, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No